CLINICAL TRIAL: NCT03580525
Title: Nicotine Delivery Rate and Its Abuse Potential: Impact of Menthol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000023289; R03DA043004-01 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Single blind, placebo-controlled, mixed-design with nicotine delivery as a within-subjects factor.
Who Masked: Participant, Investigator
Masking Description: Participant will not know nicotine dose or rate of infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- nicotine saline infusion 0.00mcg/kg/s (Experimental): 0.00 mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine saline infusion 0.00mcg/kg/s
- nicotine infusion 0.24mcg/kg/s (Experimental): 0.24mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine infusion 0.24mcg/kg/s
- nicotine infusion 0.096mcg/kg/s (Experimental): 0.096mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine infusion 0.096mcg/kg/s
- nicotine infusion 0.048mcg/kg/s (Experimental): 0.048mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine infusion 0.048 mcg/kg/s
- nicotine infusion 0.024mcg/kg/s (Experimental): 0.048mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine infusion 0.024mcg/kg/s

INTERVENTIONS:
Drug: Nicotine saline infusion 0.00mcg/kg/s — saline 0.00mcg/kg/s
  Other Names: nicotine infusion
  Arms: nicotine saline infusion 0.00mcg/kg/s
Drug: Nicotine infusion 0.24mcg/kg/s — nicotine 0.24mcg/kg/s
  Other Names: nicotine infusion
  Arms: nicotine infusion 0.24mcg/kg/s
Drug: Nicotine infusion 0.096mcg/kg/s — nicotine 0.096mcg/kg/s
  Other Names: nicotine infusion
  Arms: nicotine infusion 0.096mcg/kg/s
Drug: Nicotine infusion 0.048 mcg/kg/s — nicotine 0.048mcg/kg/s
  Other Names: nicotine infusion
  Arms: nicotine infusion 0.048mcg/kg/s
Drug: Nicotine infusion 0.024mcg/kg/s — nicotine 0.024mcg/kg/s
  Other Names: nicotine infusion
  Arms: nicotine infusion 0.024mcg/kg/s

SUMMARY:
A placebo-controlled study to enroll male and female tobacco smokers who will participate in five experimental sessions. subjects will be given an IV infusion of either saline or 1 mg nicotine at rapid, moderate or slow infusion rates (nicotine at 0.24,0.096, 0.048 and 0.024, mcg per kg body weight per sec).

DETAILED DESCRIPTION:
A placebo-controlled study that will enroll male and female tobacco smokers' menthol to participate in five experimental sessions. During the experimental session, subjects will be given an IV infusion of either saline or 1 mg nicotine at rapid, moderate or slow infusion rates (nicotine at 0.24,0.096, 0.048 and 0.024, mcg per kg body weight per sec). The infusion conditions for each experimental session will be determined in random order. Aim 1 is to establish a dose-effect curve for positive subjective effects (drug liking and good drug effects) and alleviation of smoking urges, as a function of nicotine delivery rate in menthol and non-menthol cigarette preferring smokers Aim 2 is to establish a dose-effect curve positive subjective effects and alleviation of smoking urges as a function of nicotine delivery rate. Aim 3 is to establish a dose-effect curve for nicotine's effect to alleviate symptoms of nicotine withdrawal in abstinent smokers as a function of nicotine delivery rate. Aim 4 is to establish a dose-effect curve for nicotine's acute cardiovascular health effects. Data from this project will help to establish benchmark values for nicotine's threshold effects that will guide policies on the nicotine yield of tobacco products. Presented is the time frame at which the peak change was strongest by treatment arm. The possible peak numbers could be 1, 3, 5, 7 and 10 minutes."

ELIGIBILITY:
Inclusion criteria:

* Female and male smokers, aged 18 to 35 years, who have been smoking tobacco cigarettes for at least a year
* Smoke ≥ 5 and less than 20 cigarettes per day;
* Urine cotinine levels > 100 ng/mL consistent with nicotine intake of an active smoker (23)
* Not seeking treatment at the time of the study for nicotine dependence;
* In good health as verified by medical history, screening examination, and screening laboratory tests
* For women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion criteria:

* History of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the subject to be in the study
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
* Current alcohol or substance dependence for any other recreational or prescription drugs other than nicotine
* Use of e-cigarettes more than 10 days in the past 30 days
* Urine drug screening indicating recent illicit drugs use (with the exception of marijuana).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Professor of Psychiatry
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 24 subjects were randomized, yet two subjects didn't complete all five days. Therefore, some conditions have 23 participants, and some have 22.
Groups:
- Randomized Participants: Each participant was randomized to each condition, the order and number of groups presents difficulty in the breakdown, so the number that experienced each level of the intervention is reported.
Period: Overall Study
Arm/Group | Randomized Participants
Started | 23
Nicotine Saline Infusion 0.00mcg/kg/s | 22
Nicotine Infusion 0.24mcg/kg/s | 23
Nicotine Infusion 0.096mcg/kg/s | 23
Nicotine Infusion 0.048mcg/kg/s | 22
Nicotine Infusion 0.024mcg/kg/s | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Baseline characteristics of all participants prior to randomization.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two females only completed certain days not true completers but were added to the analysis
  years | 28.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 14
  White | 7
  Native American | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Peak Changes on Items of the Drug Effects Questionnaire (DEQ) - Stimulatory Effects
Description: The peak change in the intensity of subjective effects as measured by the DEQ: Drug stimulatory effects questionnaire; Eleven questions with a minimum score of 0 to a maximum score of 100. Presented is the DEQ score at which the peak change was strongest by treatment arm. Each session took approximately 60 minutes, however the measures were only collected up to 10 minutes post infusion. This correction to the outcome time frame was made when the results were entered. Data were collected at 1, 3, 5, 7 and 10 minute intervals. The outcome measure title DEQ Stimulatory Effects measure was also updated.
Time Frame: up to 10 minutes
Population: Intention to treat analysis.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Randomized Participants: Each participant received each level of the intervention in a random order.
Arm/Group | Randomized Participants
Number analyzed (Participants) | 23
score on a scale
  nicotine saline infusion 0.00mcg/kg/s: number analyzed (Participants) | 22
  nicotine saline infusion 0.00mcg/kg/s | 7.03 (5.34)
  nicotine infusion 0.24mcg/kg/s | 37.48 (5.14)
  nicotine infusion 0.096mcg/kg/s | 41.91 (5.15)
  nicotine infusion 0.048mcg/kg/s: number analyzed (Participants) | 22
  nicotine infusion 0.048mcg/kg/s | 28.22 (5.22)
  nicotine infusion 0.024mcg/kg/s | 22.12 (5.05)

2. Primary Outcome: Peak Changes on Items of the Drug Effects Questionnaire (DEQ) - Pleasurable Effects
Description: The peak change in the intensity of subjective effects as measured by the DEQ: Drug pleasurable effects questionnaire; Eleven questions with a minimum score of 0 to a maximum score of 100. Presented is the DEQ score at which the peak change was strongest by treatment arm. Each session took approximately 60 minutes, however the measures were only collected up to 10 minutes post infusion. This correction to the outcome time frame was made when the results were entered. Data were collected at 1, 3, 5, 7 and 10 minute intervals. The outcome measure title DEQ Stimulatory Effects measure was also updated.
Time Frame: up to 10 minutes post infusion
Population: Intention to treat analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Randomized Participants
Number analyzed (Participants) | 23
score on a scale
  nicotine saline infusion 0.00mcg/kg/s: number analyzed (Participants) | 22
  nicotine saline infusion 0.00mcg/kg/s | 8.83 (5.09)
  nicotine infusion 0.24mcg/kg/s | 30.36 (4.96)
  nicotine infusion 0.096mcg/kg/s | 36.73 (4.97)
  nicotine infusion 0.048mcg/kg/s: number analyzed (Participants) | 22
  nicotine infusion 0.048mcg/kg/s | 26 (5)
  nicotine infusion 0.024mcg/kg/s | 21.19 (4.89)

ADVERSE EVENTS:
Time Frame: Up to 10 minutes post-infusion.
Arm/Group | Nicotine Saline Infusion 0.00mcg/kg/s | Nicotine Infusion 0.24mcg/kg/s | Nicotine Infusion 0.096mcg/kg/s | Nicotine Infusion 0.048mcg/kg/s | Nicotine Infusion 0.024mcg/kg/s
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/23 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23 | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03580525/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03580525/ICF_001.pdf